CLINICAL TRIAL: NCT03680261
Title: Phase III Multicenter Randomized Controlled Trial of Adjuvant Chemoradiotherapy vs Chemotherapy for Radical Resected Advanced Gastric Carcinoma Concurrent With Lymph Node Metastasis and Lymphovascular Invasion
Brief Title: Enriched-CRT 2017: Advanced Gastric Cancer With LN+ and LVI+, Chemotherapy vs. Chemoradiotherapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Xuefei.Wang, Clinical Professor,Department of General Surgery, Zhongshan Hospital, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZSGC-004
Record Dates: First submitted 2018-09-19; First posted 2018-09-21 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-09

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; Chemoradiotherapy; Chemotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Chemoradiotherapy; Drug Therapy; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adjuvant chemoradiotherapy group (Experimental): Adjuvant chemoradiotherapy (1 cycle CT: Oxaliplatin plus capecitabine (Xelox) or S-1 plus oxaliplatin (SOX), Q21d×1, Followed by RT: 45 Gray (Gy), 5d/week×5 with capecitabine or S1, Followed by 3 cycles CT: Xelox or SOX, Q21d×3) for patients enrolled in this group.
  Interventions: Radiation: chemoradiotherapy
- Adjuvant chemotherapy group (Active Comparator): Adjuvant chemotherapy (6 cycles CT: Xelox or SOX, Q21d×3) for patients enrolled in this group.
  Interventions: Drug: chemotherapy

INTERVENTIONS:
Radiation: chemoradiotherapy — CRT (1 cycle CT: Xelox or SOX, Q21d×1, Followed by RT: 45 Gray (Gy), 5d/week×5 with capecitabine or S1, Followed by 3 cycles CT: Xelox or SOX, Q21d×3) will be applied to radical resected advanced gastric cancer patients with lymph node metastasis and lymphovascular Invasion.
  Other Names: Study group (CRT)
  Arms: Adjuvant chemoradiotherapy group
Drug: chemotherapy — CT (6 cycles CT: Xelox or SOX, Q21d×3) will be applied to radical resected advanced gastric cancer patients with lymph node metastasis and lymphovascular Invasion.
  Other Names: Control group (CT)
  Arms: Adjuvant chemotherapy group

SUMMARY:
This Enriched-CRT 2017 trial is a prospective, multicenter trial for adjuvant chemoradiotherapy (CRT) and chemotherapy (CT) in radical resected advanced gastric cancer (GC) patients with lymph node metastasis (LN+) and lymphovascular Invasion (LVI+). The primary purpose of this study is to evaluate the 3-year overall survival (OS) of enrolled patients receiving adjuvant chemoradiotherapy compared with those receiving adjuvant chemotherapy. The second purpose is to evaluate 3-year disease free survival (DFS) and determine the safety of CRT compared with CT in the patients enrolled in this study.

DETAILED DESCRIPTION:
Gastric cancer is an important health problem, being the fourth most common cancer and the third leading cause of cancer-related death worldwide. Age standardized mortality rates for gastric cancer are 14.3 per 100 000 in men and 6.9 per 100 000 in women. More than 679 000 new cases and 498,000 deaths occur every year in China.

Local recurrence is considered as the most common way of recurrence for advanced gastric cancer, as well as an important factor for poor prognosis. Radiotherapy is a widely used technique in Western countries, and has been identified to have a significant role in decreasing local recurrence rate in breast cancer, and colon rectal cancer. At this moment, several randomized controlled trials have been conducted to identify the role of radiotherapy in advanced gastric cancer. Although the results from Europe (INT-0116), Dutch (CRITICS), and Korea (ARTIST) did not find that radiotherapy could improve the overall survival of enrolled patients, the sub-group analyses demonstrated that radiotherapy could improve the disease-free survival in patients with lymph node metastasis. We also found that adjuvant chemoradiotherapy could improve the survival of patients with lymph node metastasis or lymphovascular Invasion based on a large cohort study from National Cancer Database.

Therefore, our hypothesis is that advanced gastric cancer patients with lymph node metastasis or lymphovascular invasion are the group entity that could benefit from radiotherapy. At present, a new clinical trial (ARTIST II), aiming at advanced gastric cancer with positive lymph node metastasis, has been launched. China is one of the countries with the highest incidence of gastric cancer, sand nearly 80% of patients are diagnosed with advanced stage. So it's necessary to conduct the clinical research on this issue.

This Enriched-CRT 2017 trial is a prospective, multicenter trial for adjuvant chemoradiotherapy (CRT) and chemotherapy (CT) in radical resected advanced gastric cancer patients with lymph node metastasis and lymphovascular Invasion. The primary purpose of this study is to evaluate the 3-year overall survival (OS), and the second purpose is to evaluate 3-year disease free survival (DFS) and determine the safety of CRT compared with CT in the patients enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged 18-75 years；
* 2. Primary lesion is pathologically diagnosed as gastric adenocarcinoma (including Esophagogastric Junction adenocarcinoma), such as papillary adenocarcinoma, tubular adenocarcinoma, mucinous adenocarcinoma, poorly cohesive carcinoma (including signet ring cell carcinoma and other variants), and mixed adenocarcinoma;
* 3. Received radical resection: R0 gastrectomy with D1/D2 lymphadenectomy (at least 15 lymph nodes were examined);
* 4. Pathological stage pT2-4aN1-3M0 (According to American Joint Committee on Cancer (AJCC)-7th Tumor-Node-Metastasis (TNM) staging system), and with lymphovascular invasion, (LVI+);
* 5. No evidence of distant metastases was observed by perioperative imaging;
* 6. Postoperative performance status (ECOG, Eastern Cooperative Oncology Group) of 0-2;
* 7. No prior treatment of chemotherapy, radiotherapy, targeted therapy, immunotherapy, etc.;
* 8. Adequate hematological function: Hemoglobin (Hb) ≥100g/L, Neutrophil count (ANC) ≥1.5×109/L, Platelet count (PLC) ≥100×109/L;
* 9. Adequate liver function: ALT、AST ≤2.5x upper limit of normal (ULN), Alkaline phosphatase (ALP) ≤2.5x ULN, Serum total bilirubin (TBIL) <1.5x ULN, Serum albumin(Alb) ≥30g/L;
* 10. Adequate renal function: Serum creatinine ≤1.5mg/dl;
* 11. Be able of oral feeding;
* 12. Written informed consent.

Exclusion Criteria:

* 1. Synchronous or metachronous (within 5 years) malignancies;
* 2. Body temperature ≥ 38℃ or infectious disease with a systemic therapy indicated;
* 3. Severe neurological or mental disease, including seizures or dementia, which may interfere compliance and sign of consent inform.
* 4. Severe heart disease, including unstable angina pectoris, New York Heart Association (NYHA) class II or more advanced heart failure, severe arrhythmia despite medicinal treatment, or history of myocardial infarction within 12 months;
* 5. Severe respiratory disease;
* 6. Moderate or severe renal dysfunction: Creatinine clearance rate (CCR) ≤50 ml/min, or Serum creatinine >ULN ;
* 7. Upper gastrointestinal tract obstruction, physiological dysfunction, or malabsorption syndrome, which affect the absorption of oral drugs;
* 8. Peripheral nervous disease (NCI CTC version> 1.0 grade), except for patients with ony disappeared deep tendinous reflect (DTR);
* 9. Women during pregnancy or breast-feeding;
* 10. Fertile women with a positive pregnancy test, or no pregnancy test; postmenopausal within 12 months;
* 11. Fertile men or women who refuse to use contraception during the study period;
* 12. Patients are participating or have participated in another clinical trial (within 6 months);
* 13. Continuous systemic steroid therapy within 1 month (except for topical use), or received organ transplantation that needs immunosuppressive agent;
* 14. Dihydropyrimidine dehydrogenase (DPD) deficiency;
* 15. Allergy to platinum compound, or any component of drugs used in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 556 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
3-year Overall Survival | 3-year
  3-year Overall survival (OS) was defined as the time from the date of enrollment to the date of death or last visit.

SECONDARY OUTCOMES:
3-year Disease Free Survival | 3-year
  3-year Disease Free Survival (DFS) was defined as time from the date of enrollment to the date of recurrence or last visit.
Adverse effect (Safety and Tolerability) | 30 days
  The evaluation of adverse effect is based on the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Xuefei Wang, MD, PhD, Principal Investigator — Fudan University
Locations (1):
- ZhongShan hospital FuDan university, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Macdonald JS, Smalley SR, Benedetti J, Hundahl SA, Estes NC, Stemmermann GN, Haller DG, Ajani JA, Gunderson LL, Jessup JM, Martenson JA. Chemoradiotherapy after surgery compared with surgery alone for adenocarcinoma of the stomach or gastroesophageal junction. N Engl J Med. 2001 Sep 6;345(10):725-30. doi: 10.1056/NEJMoa010187. PMID 11547741
- [Background] Cunningham D, Allum WH, Stenning SP, Thompson JN, Van de Velde CJ, Nicolson M, Scarffe JH, Lofts FJ, Falk SJ, Iveson TJ, Smith DB, Langley RE, Verma M, Weeden S, Chua YJ, MAGIC Trial Participants. Perioperative chemotherapy versus surgery alone for resectable gastroesophageal cancer. N Engl J Med. 2006 Jul 6;355(1):11-20. doi: 10.1056/NEJMoa055531. PMID 16822992
- [Background] Smalley SR, Benedetti JK, Haller DG, Hundahl SA, Estes NC, Ajani JA, Gunderson LL, Goldman B, Martenson JA, Jessup JM, Stemmermann GN, Blanke CD, Macdonald JS. Updated analysis of SWOG-directed intergroup study 0116: a phase III trial of adjuvant radiochemotherapy versus observation after curative gastric cancer resection. J Clin Oncol. 2012 Jul 1;30(19):2327-33. doi: 10.1200/JCO.2011.36.7136. Epub 2012 May 14. PMID 22585691
- [Background] Sakuramoto S, Sasako M, Yamaguchi T, Kinoshita T, Fujii M, Nashimoto A, Furukawa H, Nakajima T, Ohashi Y, Imamura H, Higashino M, Yamamura Y, Kurita A, Arai K; ACTS-GC Group. Adjuvant chemotherapy for gastric cancer with S-1, an oral fluoropyrimidine. N Engl J Med. 2007 Nov 1;357(18):1810-20. doi: 10.1056/NEJMoa072252. PMID 17978289
- [Background] Ashraf N, Hoffe S, Kim R. Adjuvant treatment for gastric cancer: chemotherapy versus radiation. Oncologist. 2013;18(9):1013-21. doi: 10.1634/theoncologist.2012-0462. Epub 2013 Aug 21. PMID 23966224
- [Background] Lee J, Lim DH, Kim S, Park SH, Park JO, Park YS, Lim HY, Choi MG, Sohn TS, Noh JH, Bae JM, Ahn YC, Sohn I, Jung SH, Park CK, Kim KM, Kang WK. Phase III trial comparing capecitabine plus cisplatin versus capecitabine plus cisplatin with concurrent capecitabine radiotherapy in completely resected gastric cancer with D2 lymph node dissection: the ARTIST trial. J Clin Oncol. 2012 Jan 20;30(3):268-73. doi: 10.1200/JCO.2011.39.1953. Epub 2011 Dec 19. PMID 22184384
- [Background] Park SH, Sohn TS, Lee J, Lim DH, Hong ME, Kim KM, Sohn I, Jung SH, Choi MG, Lee JH, Bae JM, Kim S, Kim ST, Park JO, Park YS, Lim HY, Kang WK. Phase III Trial to Compare Adjuvant Chemotherapy With Capecitabine and Cisplatin Versus Concurrent Chemoradiotherapy in Gastric Cancer: Final Report of the Adjuvant Chemoradiotherapy in Stomach Tumors Trial, Including Survival and Subset Analyses. J Clin Oncol. 2015 Oct 1;33(28):3130-6. doi: 10.1200/JCO.2014.58.3930. Epub 2015 Jan 5. PMID 25559811
- [Background] Mamon HJ, Tepper JE. Combination chemoradiation therapy: the whole is more than the sum of the parts. J Clin Oncol. 2014 Feb 10;32(5):367-9. doi: 10.1200/JCO.2013.54.3108. Epub 2014 Jan 13. No abstract available. PMID 24419110
- [Background] Fisher B, Anderson S, Bryant J, Margolese RG, Deutsch M, Fisher ER, Jeong JH, Wolmark N. Twenty-year follow-up of a randomized trial comparing total mastectomy, lumpectomy, and lumpectomy plus irradiation for the treatment of invasive breast cancer. N Engl J Med. 2002 Oct 17;347(16):1233-41. doi: 10.1056/NEJMoa022152. PMID 12393820
- [Background] Wolmark N, Wieand HS, Hyams DM, Colangelo L, Dimitrov NV, Romond EH, Wexler M, Prager D, Cruz AB Jr, Gordon PH, Petrelli NJ, Deutsch M, Mamounas E, Wickerham DL, Fisher ER, Rockette H, Fisher B. Randomized trial of postoperative adjuvant chemotherapy with or without radiotherapy for carcinoma of the rectum: National Surgical Adjuvant Breast and Bowel Project Protocol R-02. J Natl Cancer Inst. 2000 Mar 1;92(5):388-96. doi: 10.1093/jnci/92.5.388. PMID 10699069
- [Background] D'Angelica M, Gonen M, Brennan MF, Turnbull AD, Bains M, Karpeh MS. Patterns of initial recurrence in completely resected gastric adenocarcinoma. Ann Surg. 2004 Nov;240(5):808-16. doi: 10.1097/01.sla.0000143245.28656.15. PMID 15492562
- [Background] Bang YJ, Kim YW, Yang HK, Chung HC, Park YK, Lee KH, Lee KW, Kim YH, Noh SI, Cho JY, Mok YJ, Kim YH, Ji J, Yeh TS, Button P, Sirzen F, Noh SH; CLASSIC trial investigators. Adjuvant capecitabine and oxaliplatin for gastric cancer after D2 gastrectomy (CLASSIC): a phase 3 open-label, randomised controlled trial. Lancet. 2012 Jan 28;379(9813):315-21. doi: 10.1016/S0140-6736(11)61873-4. Epub 2012 Jan 7. PMID 22226517
- [Background] Noh SH, Park SR, Yang HK, Chung HC, Chung IJ, Kim SW, Kim HH, Choi JH, Kim HK, Yu W, Lee JI, Shin DB, Ji J, Chen JS, Lim Y, Ha S, Bang YJ; CLASSIC trial investigators. Adjuvant capecitabine plus oxaliplatin for gastric cancer after D2 gastrectomy (CLASSIC): 5-year follow-up of an open-label, randomised phase 3 trial. Lancet Oncol. 2014 Nov;15(12):1389-96. doi: 10.1016/S1470-2045(14)70473-5. Epub 2014 Oct 15. PMID 25439693
- [Background] Songun I, Putter H, Kranenbarg EM, Sasako M, van de Velde CJ. Surgical treatment of gastric cancer: 15-year follow-up results of the randomised nationwide Dutch D1D2 trial. Lancet Oncol. 2010 May;11(5):439-49. doi: 10.1016/S1470-2045(10)70070-X. Epub 2010 Apr 19. PMID 20409751
- [Background] Li P, He HQ, Zhu CM, Ling YH, Hu WM, Zhang XK, Luo RZ, Yun JP, Xie D, Li YF, Cai MY. The prognostic significance of lymphovascular invasion in patients with resectable gastric cancer: a large retrospective study from Southern China. BMC Cancer. 2015 May 7;15:370. doi: 10.1186/s12885-015-1370-2. PMID 25947284
- [Background] Dicken BJ, Graham K, Hamilton SM, Andrews S, Lai R, Listgarten J, Jhangri GS, Saunders LD, Damaraju S, Cass C. Lymphovascular invasion is associated with poor survival in gastric cancer: an application of gene-expression and tissue array techniques. Ann Surg. 2006 Jan;243(1):64-73. doi: 10.1097/01.sla.0000194087.96582.3e. PMID 16371738
- [Background] Lee JH, Kim MG, Jung MS, Kwon SJ. Prognostic significance of lymphovascular invasion in node-negative gastric cancer. World J Surg. 2015 Mar;39(3):732-9. doi: 10.1007/s00268-014-2846-y. PMID 25376868
- [Background] Dikken JL, van Sandick JW, Maurits Swellengrebel HA, Lind PA, Putter H, Jansen EP, Boot H, van Grieken NC, van de Velde CJ, Verheij M, Cats A. Neo-adjuvant chemotherapy followed by surgery and chemotherapy or by surgery and chemoradiotherapy for patients with resectable gastric cancer (CRITICS). BMC Cancer. 2011 Aug 2;11:329. doi: 10.1186/1471-2407-11-329. PMID 21810227